CLINICAL TRIAL: NCT03902600
Title: Moderately Hypofractionated Photon and Proton Chemoradiotherapy as Definitive or Neoadjuvant Therapy in Non-metastatic Pancreas Cancer With Assessment of Treatment Response Utilizing Molecular Biomarkers
Brief Title: A Study of Photon and Proton Chemoradiotherapy as Definitive or Neoadjuvant Therapy in Non-Metastatic Pancreatic Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ROR1741; NCI-2021-13899 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); ROR1741 (Other: Mayo Clinic Radiation Oncology); 17-011198 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Moderately Hypofractionated RT — Patients will be treated with moderately hypofractionated radiation treatment

SUMMARY:
This study will observe side effects for patients who receive a 3-week course of radiation and chemotherapy for pancreas cancer. Blood samples will be collected before and after treatment to assess pancreas cancer DNA levels and its impact on outcomes.

ELIGIBILITY:
Inclusion Criteria: -Age ≥ 18 years

* Histological confirmation of adenocarcinoma of the pancreas (head, body, or tail of pancreas)
* Imaging consistent with T1-4, N0-2, M0 pancreas cancer, including potentially resectable, borderline resectable, or unresectable disease as per National Comprehensive Cancer Network (NCCN) classification. When CT of the chest, abdomen, and pelvis are performed, this must be with contras per pancreas protocol. Imagining with positron emission tomography (PET)/magnetic resonance imaging (MRI) alone is acceptable on study. If PET/CT is performed, a separate pancreas protocol CT is required for inclusion.
* Must have received neoadjuvant chemotherapy at the discretion of medical oncology
* Medical oncology consultation to confirm that patient is an appropriate candidate for concurrent chemotherapy and surgical oncology consultation for confirmation of resection status.

  * Note: Patients who have received previous chemotherapy for pancreatic cancer are allowed to participate in this study, unless they experienced a previous allergic reaction to the drugs used in this study.
* Planned to receive CRT, consisting of proton beam therapy (PBT) or intensity-modulated radiation therapy (IMRT) (45 Gy/15 fractions) with concurrent chemotherapy with 5FU or Capecitabine.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 or Karnofsky Performance Status 70-100 (Appendix III).
* Willing to sign consent onto the Mayo Clinic Radiotherapy Patient Outcomes Registry and Biobanking study, Institutional Review Board (IRB) 15-000136

  * Patients do not need to agree to Biobank blood draw.
  * Patients at Mayo Clinic Arizona are not required to consent to the Registry.
* Willing to sign consent for blood collection onto the Pancreas SPORE, IRB 354-06.
* Able to complete standard of care clinical questionnaire(s) by themselves or with assistance.

Exclusion Criteria:

* Presence of non-regional nodal involvement or distant metastatic disease (M1)
* Prior RT to the thorax, abdomen, or pelvis
* History of prior malignancy < 2 years of enrollment, except non-melanotic skin cancer or carcinoma-in-situ of the cervix
* Immunocompromised patients and patients known to be HIV positive and not currently receiving antiretroviral therapy.

  * Note: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.
* Receiving any investigational agent concurrent with CRT which would be considered as a treatment for the primary neoplasm.
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic or psychiatric illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Acute grade 3 or higher GI AEs | Up to 3 months after CRT
  Acute grade 3 or higher gastrointestinal (GI) adverse events (AEs) possibly, probably, or definitely related to hypofractionated concurrent chemoradiotherapy (CRT)

SECONDARY OUTCOMES:
Late grade 3 or higher GI AEs | 3 months to 2 years after CRT
  Late grade 3 or higher GI AEs attributable to hypofractionated concurrent CRT
Local-regional recurrence | 2 years after CRT
  Defined as disease recurrence within the residual pancreas, anastomosis, celiac or superior mesenteric plexus, or regional lymphatic stations with or without metastatic disease, estimated from the time of registration. Metastatic disease will be defined as tumor recurrence in a distant nodal or organ site.
Progression free survival (PFS) | 2 years after CRT
  Defined as freedom from local-regional or metastatic progression or death of any cause, estimated from the time of registration.
Overall survival (OS) | 2 years after CRT or until death
  Defined as freedom from any cause of death, estimated from the time of registration.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W. Merrell, MD, Principal Investigator — Mayo Clinic in Rochester; Krishan R. Jethwa, MD, Principal Investigator — Mayo Clinic in Rochester; Terence T. Sio, MD, MS, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials